CLINICAL TRIAL: NCT04002349
Title: Study of Medication for Nonallergic Rhinitis (NAR) Based on Cluster Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Institute of Otolaryngology (Unknown); Shanghai Johnson & Johnson Pharmaceuticals, Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR-Med-NAR-Cluster
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Determination of the Efficacy of Different Medications for Idiopathic Rhinitis; Impact of Different Medications on Biomarkers of Idiopathic Rhinitis; Safety and Tolerance of Different Medications for Idiopathic Rhinitis
MeSH Terms: interventions — Budesonide; Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: Placebo group (Placebo Comparator): Treated by 0.9% Natural saline (NS) nasal spray: 2 sprays each side daily in the morning
  Interventions: Drug: 0.9% natural saline
- B: Budesonide Nasal Spray (Rhinocort) (Experimental): Treated by Budesonide Nasal Spray (Rhinocort, Shanghai Johnson & Johnson Pharmaceuticals, Ltd.) nasal spray: 2 sprays each side daily in the morning
  Interventions: Drug: Budesonide Nasal Spray (Rhinocort, Shanghai Johnson & Johnson Pharmaceuticals, Ltd.)
- C: Levocabastine Nasal Spray (Livostine) (Experimental): Treated by Levocabastine(Livostinet, Shanghai Johnson & Johnson Pharmaceuticals, Ltd.) Nasal Spray: 2 sprays each side daily in the morning
  Interventions: Drug: Levocabastine Nasal Spray (Livostine, Shanghai Johnson & Johnson Pharmaceuticals, Ltd.)
- D: Combined Treatment (Experimental): Treated by Budesonide Nasal Spray (Rhinocort, Shanghai Johnson & Johnson Pharmaceuticals, Ltd.) nasal spray: 2 sprays each side daily in the morning and Levocabastine(Livostinet, Shanghai Johnson & Johnson Pharmaceuticals, Ltd.) Nasal Spray: 2 sprays each side daily in the morning
  Interventions: Drug: Budesonide Nasal Spray (Rhinocort, Shanghai Johnson & Johnson Pharmaceuticals, Ltd.); Drug: Levocabastine Nasal Spray (Livostine, Shanghai Johnson & Johnson Pharmaceuticals, Ltd.)

INTERVENTIONS:
Drug: Budesonide Nasal Spray (Rhinocort, Shanghai Johnson & Johnson Pharmaceuticals, Ltd.) — Detailed in arm descriptions
  Arms: B: Budesonide Nasal Spray (Rhinocort); D: Combined Treatment
Drug: Levocabastine Nasal Spray (Livostine, Shanghai Johnson & Johnson Pharmaceuticals, Ltd.) — Detailed in arm descriptions
  Arms: C: Levocabastine Nasal Spray (Livostine); D: Combined Treatment
Drug: 0.9% natural saline — Detailed in arm descriptions
  Arms: A: Placebo group

SUMMARY:
Chronic rhinitis (CR) is one of the most common nasal mucosal diseases in the world. In China, about 140 million people suffer from this disease. Chronic rhinitis can lead to severe economic and social burden, as well as the potential risk of developing other chronic diseases such as asthma and chronic sinusitis. Therefore, it is of great significance to explore the classification and treatment strategies of chronic rhinitis in order to improve the health level of Chinese people.

ELIGIBILITY:
Inclusion Criteria:

* Not younger than 18 years old
* Diagnosed as idiopathic rhinitis
* Signed and volunteered for the study

Exclusion Criteria:

* Comorbid airway diseases including (but not limited to) upper airway infection, chronic rhinosinusitis, nasal polyps
* Allergic to the medicines about to study
* Having used oral glucocorticoids or antihistamine agents within 30 days of the enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Relief of bothersome symptoms | 2 weeks
  Determined by change of visual analog scale for symptoms

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Yifan Meng, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided